CLINICAL TRIAL: NCT06500104
Title: The Effects of Kefir on Pediatric Obesity
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH112-REC2-145
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kefir (Experimental): Daily oral kefir peptide (KEFPEP®) intake, dosage: 1.2 gram per day for 12 weeks
  Interventions: Dietary Supplement: Kefir peptide
- Placebo (Placebo Comparator): Daily oral glucose powder intake, dosage: 805mg per day for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Kefir peptide — Dosage: 1.2 gram kefir peptide daily oral intake for 12 weeks
  Arms: Kefir
Dietary Supplement: Placebo — Glucose powder
  Arms: Placebo

SUMMARY:
Kefir, a traditional fermented dairy product in the North Caucasus region, is produced through the fermentation of milk by lactic acid bacteria and yeast. In murine studies, it has been observed that consumption of kefir by obese mice resulted in significantly reduced body weight compared to non-kefir-consuming obese mice. Furthermore, insulin resistance and fatty liver conditions showed improvement in the kefir-fed obese mice. Kefir was found to have its effects on obesity-related conditions through the inhibition of lipid synthesis, stimulation of fatty acid oxidation, elevation of basal metabolic rate, and modulation of oxidative damage.

Obesity has emerged as a global epidemic, and its prevalence in pediatric population is rapidly increasing. Obesity is defined as having a body mass index (BMI) above the 95th percentile for the age. According to statistics from the Health Promotion Administration in Taiwan, the prevalence of obesity among elementary and junior high school students in 2021 was 27.1% and 31.2%, respectively. This implies that approximately one out of every three to four students is obese. Insulin resistance and fatty liver are two common manifestations of childhood obesity. Insulin resistance is found closely linked to type 2 diabetes. Prolonged and chronic fatty liver can progress to cirrhosis and even hepatocellular carcinoma. Effective management of obesity holds the occurrence of these diseases. The objective of this study is to analyze the potential benefits of incorporating kefir into the diet of obese children regarding the improvement of obesity-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* body weight above 40 kilograms, body mass index (BMI)-for-age above the 95th percentile

Exclusion Criteria:

* diabetes mellitus, liver diseases other than non-alcoholic fatty liver disease, cardiovascular diseases other than hypertension and dyslipidemia, renal diseases, neurologic diseases, growth hormone deficiency, thyroid diseases, adrenal disorders, any use of medication for more than 6 months before or during this study, and any adverse responses to dairy products.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-07-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
BMI | From enrollment to the end of treatment at 12 weeks
  BMI

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Children's Hospital, Taichung, Taiwan